CLINICAL TRIAL: NCT01387893
Title: Study of a Self-Administered Maneuver to Initiate and Maintain Urine Flow Impeded by Benign Prostatic Hyperplasia
Brief Title: A Self-Administered Maneuver to Relieve Symptoms Suggestive of Benign Prostatic Hyperplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CN-07PFren-01-H; 02-0115-9922 (Other Grant/Funding Number: KPNC Community Benefit Research Fund Grant #02-0115-9922)
Record Dates: First submitted 2011-06-29; First posted 2011-07-06 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia; BPH; Lower Urinary Tract Symptoms; LUTS; Self-Administered Maneuver; Symptomatic Relief; Digital Repetitive Infrapubic Pressure maneuver
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Immediate & Delayed Instruction (Experimental): Male patients with mild to moderate lower urinary tract symptoms will alternately be assigned to either immediate intervention or delayed intervention groups. Statistical assessments will be performed to establish comparability of baseline characteristics in the two groups.
  Interventions: Behavioral: the Digital Repetitive Infrapubic Pressure maneuver

INTERVENTIONS:
Behavioral: the Digital Repetitive Infrapubic Pressure maneuver — The Digital Repetitive Infrapubic Pressure maneuver is performed by exerting moderate inwards pressure with the index and middle fingers, spread slightly apart, palm-side up, pushing into the fold of skin at the base of the penis, where it comes forward beneath the pubic bones, one fingertip on each side of the penis' suspensory ligament. By repeatedly pushing inwards and slightly upwards, at a rate of about once per second, to a distance of about two centimeters, at times of significant urinary hesitancy it is often possible either to initiate spontaneous flow, or to pass a small quantity of urine with each push, such that after a minute or two one can empty the bladder to a satisfactory degree. While a few men find it useful when voiding in a standing position, for the majority, the maneuver requires a forward-leaning seated posture for optimal results.

SUMMARY:
The objective of this study was to evaluate the effectiveness of the Digital Repetitive Infrapubic Pressure maneuver, a self-administered procedure used to provide symptomatic relief in initiating and maintaining urine flow impeded by benign prostatic hyperplasia.

DETAILED DESCRIPTION:
Eligible patients were alternately assigned to either immediate instruction on the use of the Digital Repetitive Infrapubic Pressure maneuver (immediate intervention group) or to a return appointment to receive instructions in the maneuver four weeks after the initial assessment date (delayed intervention group). Patients were to utilize the procedure on every occasion they had difficulty initiating, maintaining, or completing urine flow between the time of their instruction and their subsequent visit. At the initial assessment visits and the final visit, the patients completed an International Prostate Score Sheet (IPSS). A telephone survey was conducted with all patients an average of nine months following their instruction in the maneuver, to determine the extent to which they were still using it.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate symptoms of difficulty initiating and maintaining the flow of urine
* not currently receiving treatment for the condition
* not taking an alpha-blocker at least one month before randomization
* not taking 5-alpha reductase inhibitor six months or more before randomization.

Exclusion Criteria:

* non-ambulatory
* taking medications known to affect urination,
* any of the following: a debilitating concomitant illness, a history of prostate or bladder cancer or prostate surgery or radiation treatment to the pelvis, urethral stricture, neurogenic bladder, current urinary tract infection or otherwise potentially compromised urinary tract systems, a creatinine level of over 3.0 mg per deciliter, or a residual urinary volume after voiding of over 350 cubic centimeters.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Change in the International Prostate Symptom Score (IPSS) | The initial time frame was to average four weeks. There was a subsequent follow up time frame averaging nine months
  The primary efficacy analyses compared the change over time in the IPSS scores between the immediate and the delayed intervention groups, and the changes over time between pre- and post-intervention scores for all patients completing the study.

SECONDARY OUTCOMES:
Continued use of technique following intervention | Nine months after intial 4 week intervention
  Secondary efficacy analysis: The number of patients (percentage of patients completing the study) who were still employing the technique on follow-up nine months later.

CONTACTS AND LOCATIONS:
Overall Officials: Perrin L French, MD, Principal Investigator — Kaiser Permanente Santa Clara
Locations (1):
- Kaiser Permanente, Santa Clara, California, United States